CLINICAL TRIAL: NCT06200571
Title: Characterization of the Immunological and Vascular Effects of Aspirin in Prevention of Preeclampsia in High-risk Nulliparous Women
Brief Title: Biological Changes Associated With High Risk of Preeclampsia in Nulliparous Women
Acronym: PRERISK
Status: Enrolling by invitation | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Alesund Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 537602
Record Dates: First submitted 2023-12-08; First posted 2024-01-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urin, placenta, umbilical cord blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nulliparous women with low risk for preeclampsia: Nulliparous women with low risk for preeclampsia by FMF-screening in the first trimester. Follow-up in week 22-24, 32, 36 and 6 months after delivery wtih clinical measurements, ultrasound doppler, blood- and urin samples.
- Nulliparous women with high risk for preeclampsia without aspirin: Nulliparous women with high risk for preeclampsia by FMF-screening in the first trimester. Follow-up in week 22-24, 32, 36 and 6 months after delivery wtih clinical measurements, ultrasound doppler, blood- and urin samples.
- Nulliparous women with high risk for preeclampsia with aspirin: Nulliparous women with high risk for preeclampsia by FMF-screening in the first trimester. Follow-up in week 22-24, 32, 36 and 6 months after delivery wtih clinical measurements, ultrasound doppler, blood- and urin samples. Aspirin tablets 150 mg daily in the evening from first trimester to week 36 of pregnancy.

SUMMARY:
Primary outcome

1. to identify biological changes in nulliparous women at high risk for preeclampsia defined by combined screening by Fetal Medicine Foundation (FMF)
2. to identify biological effects of aspirin in nulliparous women with high risk for preeclampsia

Secondary outcomes include findings of longitudinal development and predictive potential of biological markers associated with high-risk for preeclampsia and aspirin treatment.

The main questions it aims to answer are:

* Is high risk for preeclampsia associated with biological changes during pregnancy?
* How does aspirin modulate the biological changes associated with high risk for preeclampsia?

Nulliparous women will undergo routine clinical care at two regional hospitals with different treatment strategies, and selected to the study in three groups: low risk of preeclampsia, high risk of preeclampsia without aspirin, and high-risk of preeclampsia with aspirin treatment.

DETAILED DESCRIPTION:
St. Olavs Hospital offers FMF-screening in week 11-14 and aspirin treatment through the "Implementing Screening for Preeclampsia in Norway With Aspirin Discontinuation at 24-28 Weeks - a Randomized Controlled Trial" (NCT06108947). FMF-screening and aspirin treatment are not part of routine clinical care at Alesund Hospital according to current recommendations from the Norwegian health authorities. Alesund Hospital will therefore perform FMF-screening only to determine the project specific study groups. Researchers will compare the three groups to identify biological changes associated with high risk for preeclampsia and the effect of aspirin.

FMF- screening will be performed in week 11-14 after written, informed consent (approved by the the Regional Committee for Medical and Health Research Ethics in Central Norway (REK-midt), REK 537602). Screening includes patient history, blood pressure, uterine artery mean pulsatile index and serum placenta growth factor (PlGF). Standardized blood pressure will be measured by trained personnel. Ultrasound scans will be performed by FMF certified doctors and midwives working at Alesund Hospital and the Center for Fetal Medicine at St.Olavs Hospital in Trondheim. PlGF in maternal serum will be analyzed with Roche or Kryptor technology.

The investigators will include around 200 women, 18 years or older, with a singleton live fetus, in three groups:

* Nulliparous women with low risk for preeclampsia (at both hospitals)
* Nulliparous women with high risk for preeclampsia without aspirin (at Alesund Hospital)
* Nulliparous women with high risk for preeclampsia with aspirin (at St. Olavs Hospital)

Follow-up: all three groups will have visits in week 22-24, 32 and 38, and standard antenatal care after 37 weeks until delivery. Fetal growth and Doppler will be assessed at the scheduled visits and according to clinical judgement by obstetricians at the outpatient clinic of the hospital. Women will have follow-up 6 months after birth.

Blood and urine will be sampled at five time points for all three groups (week 11-14, 22-24, 32, 38 and 6 months after birth) for biological analyses. Placenta samples and umbilical venous blood will be sampled at delivery.

Biological materials will be investigated to answer the research questions described. Biological changes in serum will be measured as cytokines by multiplex, metabolites by NMR-analysis, and lipids by NMR-analysis. Vascular changes in the placenta will be measured by histopathological evaluation.

The study will be registered in Clinicaltrials.gov

Funding and sponsors: The study is funded by Helse-Midt Norge RHF. The funding source has played no role in design of the study and will have no role in data collection, analyses, interpretation or publication.

Participants: Ann-Charlotte Iversen, professor, Phd, Project leader Åse Turid Rossevatn Svoren, consultant, MD, Phd candidate, Kjell Åsmund Salvesen, professor, MD, PhD, Solveig Bjellmo, consultant, MD, Phd

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* nulliparous women
* singleton live fetus
* FMF risk > 1/100 (high risk), or < 1/150 (low risk)

Exclusion Criteria:

* not speaking Norwegian or English language
* fetal anomalies diagnosed with ultrasound

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female, only pregnant women
Study Population: Nulliparous women with low and high risk for preeclampsia, defined by FMF-screening in week 11-14 of pregnancy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal serum cytokine profile in week 11-13, 22-24, 32 and 38 and 6 months post partum | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Maternal serum cytokine profile in week 11-13, 22-24, 32 and 38 and 6 months post partum | December 2028
  Significant difference between high-risk pregnancies with and without aspirin

SECONDARY OUTCOMES:
Maternal serum metabolite profile in week 11-13, 22-24, 32 and 38 and 6 months post partum | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Maternal serum lipid profile in week 11-13, 22-24, 32 and 38 and 6 months post partum | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Maternal serum metabolite profile in week 11-13, 22-24, 32 and 38 and 6 months post partum | December 2028
  Significant difference between high-risk pregnancies with and without aspirin
Maternal serum lipid profile in week 11-13, 22-24, 32 and 38 and 6 months post partum | December 2028
  Significant difference between high-risk pregnancies with and without aspirin
Maternal vascular malperfusion in the placenta | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Fetal vascular malperfusion in the placenta | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Maternal vascular malperfusion in the placenta | December 2028
  Significant difference between high-risk pregnancies with and without aspirin
Fetal vascular malperfusion in the placenta | December 2028
  Significant difference between high-risk pregnancies with and without aspirin
Fetal cord serum cytokine profile | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Fetal cord serum metabolite profile | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Fetal cord serum lipid profile | December 2028
  Significant difference between low and high-risk pregnancies defined by FMF-screening
Fetal cord serum cytokine profile | December 2028
  Significant difference between high-risk pregnancies with and without aspirin
Fetal cord serum metabolite profile | December 2028
  Significant difference between high-risk pregnancies with and without aspirin
Fetal cord serum lipid profile | December 2028
  Significant difference between high-risk pregnancies with and without aspirin

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Charlotte Iversen, Professor, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Alesund Hospital, Ålesund
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
It may be necessary to include other researchers for planned analysis of the biological materials, for instance for pathological classification of placental tissue. Limited individual clinical information such as diagnosis and gestational age at delivery may be shared, but only in deidentified form.
  When publishing research findings from the project in international peer-reviewed journals, it may be required to publish individual research data along with very limited clinical information in a repository, but only in anonymized form.

REFERENCES:
- See also: Cytokine patterns in maternal serum from first trimester to term and beyond — https://doi.org/10.3389/fimmu.2021.752660
- See also: Metabolomic biomarkers in serum and urine in women with preeclampsia — https://doi.org/10.1371/journal.pone.0091923